CLINICAL TRIAL: NCT01748279
Title: The Effects of Atorvastatin Treatment in COPD Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Bialystok (Other)
Responsible Party: Principal Investigator, Robert M. Mroz, Associate Professor, Medical University of Bialystok
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 113-46-966; N N402 593440 (Other: Polish National Centre of Science)
Record Dates: First submitted 2012-12-09; First posted 2012-12-12 (Estimated); Last update posted 2013-04-23 (Estimated); Status verified 2013-04

CONDITIONS: COPD
Keywords: COPD; Atorvastatin; statins; COPD treatment; microarrays
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Atorvastatin; Formoterol Fumarate; lactitol; Lactose

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atorvastatin (Active Comparator): 40 mg of Atorvastatin once daily as add-on to Formoterol only 12 weeks therapy.
  Interventions: Drug: Atorvastatin; Drug: Formoterol
- Lactose tablet (Placebo Comparator): One tablet taken once a day as add-on treatment to Formoterol baseline 12 weeks therapy.
  Interventions: Drug: Formoterol; Drug: Lactose tablet

INTERVENTIONS:
Drug: Atorvastatin
  Other Names: Sortis 40, manufactured by Godecke GmBH Mooswaldallee 1 790900; Freiburg, Germany
  Arms: Atorvastatin
Drug: Formoterol — 12mcg of Foradil BID as maintenance COPD treatment in both treatment arms
  Other Names: Foradil, Novartis,
Drug: Lactose tablet — One lactose tablet taken once a day as add-on treatment to Formoterol therapy
  Arms: Lactose tablet

SUMMARY:
Rationale: Retrospective studies suggest that statins improve outcomes in COPD patients possibly as a result of an anti-inflammatory effect.

Objectives: To determine whether statins have an anti-inflammatory effect on the lungs of patients with COPD.

A controlled, parallel group study to compare the effects of Atorvastatin in comparison to placebo as an add-on treatment to Formoterol therapy in patients with mild to moderate COPD in group of 20 patients. All subjects will have spirometry, lung volumes, DLCO, SGRQ, 6MWD, serum lipids and hs-CRP measured before and after treatment. Bronchoscopy and transbronchial lung biopsy (TBB) will be carried out at baseline and after 12 weeks of treatment, and TBB specimens will be processed for histology, immunohistochemistry and microarray analysis.

ELIGIBILITY:
Inclusion Criteria:

. Written informed consent must be obtained before any assessment is performed. 2. Male and female adults aged ≥40 years, who have signed an Informed Consent Form prior to initiation of any study-related procedure.

3. Patients with moderate to very severe stable COPD (Stage II-IV) according to the GOLD guidelines.

4. Patients with a post-bronchodilator FEV1 < 80% of the predicted normal, and a post-bronchodilator FEV1/FVC < 0.70 at Visit 1.

5. Current or ex-smokers who have a smoking history of at least 10 pack years

Exclusion criteria

1. Pregnant or nursing (lactating) women
2. Women of child-bearing potential, unless they are using effective methods of contraception during dosing of study treatment. 5. 3. Patients with a clinically significant abnormality at Visit 1.

4. Patients with a clinically relevant laboratory abnormality at Visit 1 5. Patients with a history of malignancy of any organ system (including lung cancer).

6. Patients contraindicated for treatment with statins 7. Patients unable to perform acceptable spirometry and lung volumes procedures.

8. Patients who have had a COPD exacerbation that required treatment with antibiotics and/or oral corticosteroids and/or hospitalization in the 6 weeks prior to Visit 1.

9. Patients who have had a respiratory tract infection within 4 weeks prior to Visit 1.

10. Patients requiring oxygen therapy (>15 hr/day) on a daily basis for chronic hypoxemia 11. Patients with any history of asthma or onset of symptoms prior to age 40 years.

12. Patients with concomitant pulmonary disease, (e.g. lung fibrosis, sarcoidosis, interstitial lung disease, pulmonary hypertension, tuberculosis).

13. Patients with primary bronchiectasis. 14. Patients with a diagnosis of α-1 anti-trypsin deficiency. 15. Patients with pulmonary lobectomy or lung volume reduction surgery or lung transplantation.

16. Patients participating in or planning to participate in the active phase of a supervised pulmonary rehabilitation program during the study.

17. Patients receiving any medications in the class listed in Table 5.1 18. Use of other investigational drugs within 30 days prior to visit 1.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-12; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Change in CD45+ cells expression over study period | 12 weeks
  Change in CD45+ cells expression measured by immunohistochemistry in lung biopsy samples assessed before and after 12 weeks of treatment
Change in gene expression over study period | 12 weeks
  Change in gene expression measured in lung biopsy samples measured using microarrays before and after 12 weeks of treatment

SECONDARY OUTCOMES:
Change in health related quality of life over study period | 12 weeks
  Change in health related quality of life assessed by St. George's respiratory questionnaire before and after 12 weeks of treatment
Change in 6-Minute Walk Distance over study period | 12 weeks
  Change in 6-Minute Walk Distance measured according to 6-MWD protocol before and after 12 weeks of treatment
Change in intimal-medial thickness over study period | 12 weeks
  Change in intimal-medial thickness (IMT) measured in the common carotid artery (CCA) using a standard technique.
Change in hs-CRP over study period | 12 weeks
  Change in serum hs-C-reactive protein (hs-CRP) measured before and after 12 weeks of therapy
Change in total cholesterol, LDL and HDL-Cholesterol and triglycerides over study period | 12 weeks
  Change in total cholesterol, LDL and HDL-Cholesterol, and triglycerides measured before an after 12 weeks of therapy.

OTHER OUTCOMES:
Change in lung volumes over study period | 12 weeks
  Change in lung volumes measured using body plethysmography before and after 12 weeks of treatment
Change in FEV1 over study period | 12 weeks
  Change in FEV1 measured using spirometry before and after 12 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Mroz, MD, Principal Investigator — Medical University of Bialystok, Bialystok, Poland
Locations (1):
- Department of Lung Diseases and Tuberculosis, Medical University of Bialystok, Bialystok, Poland

REFERENCES:
- [Derived] Mroz RM, Lisowski P, Tycinska A, Bierla J, Trzeciak PZ, Minarowski L, Milewski R, Lisowska A, Boros P, Sobkowicz B, Duszewska AM, Chyczewska E, Musial WJ, MacNee W. Anti-inflammatory effects of atorvastatin treatment in chronic obstructive pulmonary disease. A controlled pilot study. J Physiol Pharmacol. 2015 Feb;66(1):111-28. PMID 25716971